CLINICAL TRIAL: NCT01719653
Title: A Randomized Comparison of Five Low Volume Bowel Preparations for Colonoscopy
Brief Title: A Comparison of 5 Low Volume Bowel Preparations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gastroenterology Services, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1220121180
Record Dates: First submitted 2012-10-28; First posted 2012-11-01 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: Colonoscopy; Bowel Preparation; MiraLAX; Gatorade; PEG-3350; MoviPrep; SUPREP; Chicago Bowel Preparation Scale; Boston Bowel Preparation Scale
MeSH Terms: interventions — polyethylene glycol 3350; gatorade; MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MiraLAX 306 g (Day-Prior) (Active Comparator): MiraLAX 306 g and Gatorade 64 oz (1/2 gallon) consumed the day-prior to the colonoscopy as follows: Miralax 51 g at 12 noon; Gatorade 64 oz mixed with Miralax 255 g from about 6 PM to 9 PM
  Interventions: Drug: MiraLAX; Other: Gatorade
- MiraLAX 357 g (Day-Prior) (Experimental): MiraLAX 357 g and Gatorade 64 oz (1/2 gallon) consumed the day-prior to the colonoscopy as follows: Miralax 68 g at 12 noon; Gatorade 64 oz mixed with Miralax 289 g from about 6 PM to 9 PM.
  Interventions: Drug: MiraLAX; Other: Gatorade
- MiraLAX 306 g (Split-Dose) (Experimental): MiraLAX 306 g and Gatorade 64 oz (1/2 gallon) consumed as a split-dose as follows: Gatorade 32oz mixed with Miralax 153 g from about 6 PM to 8 PM the day prior to the colonoscopy; Gatorade 32oz mixed with Miralax 153 g from about 2-4 hours prior to the colonoscopy.
  Interventions: Drug: MiraLAX; Other: Gatorade
- MoviPrep (Split-Dose) (Active Comparator): MoviPrep consumed as a split-dose as follows: MoviPrep 1 liter consumed from about 6 PM to 7 PM the day prior to the colonoscopy followed by 0.5 liter of clear liquids; MoviPrep 1 liter consumed from 3-4 hours prior to the colonoscopy followed by 0.5 liter of clear liquids.
  Interventions: Drug: MoviPrep
- SUPREP (Split-Dose) (Active Comparator): SUPREP consumed as a split-dose as follows: SUPREP 16 oz consumed from about 6 PM to 7 PM the day prior to the colonoscopy followed by 32 oz of clear liquids; SUPREP 16 oz consumed from 3-4 hours prior to the colonoscopy followed by 32 oz of clear liquids.
  Interventions: Drug: SUPREP

INTERVENTIONS:
Drug: MiraLAX — MiraLAX consumed as described in each arm.
  Other Names: PEG-3350
  Arms: MiraLAX 306 g (Day-Prior); MiraLAX 306 g (Split-Dose); MiraLAX 357 g (Day-Prior)
Other: Gatorade — Gatorade consumed as described in each arm.
  Arms: MiraLAX 306 g (Day-Prior); MiraLAX 306 g (Split-Dose); MiraLAX 357 g (Day-Prior)
Drug: MoviPrep — MoviPrep consumed as described in each arm.
  Arms: MoviPrep (Split-Dose)
Drug: SUPREP — SUPREP consumed as described in each arm.
  Arms: SUPREP (Split-Dose)

SUMMARY:
The purpose of this investigation is to compare 3 versions of MiraLAX/Gatorade, MoviPrep and SUPREP to see which preparation cleanses the colon best and which preparation is best tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old planning to undergo an elective colonoscopy will be eligible for inclusion in our study. We would prefer to exclude as few groups as possible since in clinical practice these less well studied groups often need a colonoscopy and will need to have a colonoscopy preparation.

Exclusion Criteria:

1. Patients who are allergic (this is very rare) or intolerant to any of the study drugs.
2. Patients who are pregnant.
3. Patients who required multiple day colon preparations (2 days prior and 1 day prior) in the past will be excluded.
4. Patients with ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or toxic megacolon would not be considered elective colonoscopies and are excluded.
5. Patients with known renal disease (baseline creatinine greater than 1.50 mg/dl) will need to be excluded due to the magnesium in SUPREP which is contraindicated in patients with significant renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1079 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gerard, MD, Principal Investigator — Gastroenterology Services, Ltd.
Locations (1):
- Gastroenterology Services, Downers Grove, Illinois, United States

REFERENCES:
- [Result] Gerard DP, Foster DB, Holden JL, Kang J, Raiser MW. Clinical Trial of 1000 Subjects Randomized to 5 Low-Volume Bowel Preparations for Colonoscopy and Their Acceptance of Split-Dose Bowel Preparations. J Clin Gastroenterol. 2017 Jul;51(6):512-521. doi: 10.1097/MCG.0000000000000575. PMID 27433812

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MiraLAX 306 g (Day-Prior) | MiraLAX 357 g (Day-Prior) | MiraLAX 306 g (Split-Dose) | MoviPrep (Split-Dose) | SUPREP (Split-Dose)
Started | 209 | 213 | 218 | 218 | 221
Completed | 200 | 200 | 200 | 200 | 200
Not Completed | 9 | 13 | 18 | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MiraLAX 306 g (Day-Prior) | MiraLAX 357 g (Day-Prior) | MiraLAX 306 g (Split-Dose) | MoviPrep (Split-Dose) | SUPREP (Split-Dose) | Total
Number analyzed (Participants) | 200 | 200 | 200 | 200 | 200 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (12.7) | 61.3 (12.4) | 59.1 (11.3) | 60.1 (11.4) | 60.6 (11.2) | 60.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 99 | 101 | 97 | 99 | 495
  Male | 101 | 101 | 99 | 103 | 101 | 505
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 200 | 200 | 200 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Chicago Bowel Preparation Scale
Description: The quality of the colon preparation as graded using our new Chicago Bowel Preparation Scale (BPS) (Adventist Midwest Region Institutional Review Board, AMH 2010-01-80; ClinicalTrials.gov NCT01063049). Chicago BPS total score is ranges from 0 (very poor) to 36 (outstanding). Modified Chicago BPS total score is ranges from 0 (very poor) to 33 (outstanding). Chicago BPS Fluid score is ranges from 0 (dry) to 3 (wet).
Time Frame: At completion of colonoscopy - day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MiraLAX 306 g (Day-Prior) | MiraLAX 357 g (Day-Prior) | MiraLAX 306 g (Split-Dose) | MoviPrep (Split-Dose) | SUPREP (Split-Dose)
Number analyzed (Participants) | 200 | 200 | 200 | 200 | 200
units on a scale
  Chicago BPS Total Score | 33.54 (4.28) | 34.00 (4.25) | 34.67 (3.58) | 34.95 (3.39) | 35.16 (2.34)
  Modified Chicago BPS Total Score | 31.82 (3.59) | 32.14 (3.69) | 32.33 (2.93) | 32.54 (2.92) | 32.65 (1.72)
  Chicago BPS Fluid Score | 0.90 (0.83) | 1.03 (0.89) | 1.84 (0.90) | 1.45 (0.82) | 1.30 (0.91)
Statistical Analysis 1: Comparison: MiraLAX 306 g (Day-Prior) vs MiraLAX 357 g (Day-Prior) vs MiraLAX 306 g (Split-Dose) vs MoviPrep (Split-Dose) vs SUPREP (Split-Dose); All 5 arms were compared pair-wise. 1=G+PEG-306 2=G+PEG-357 3=G+PEG-Split 4=PEG+Asc-Split 5=SS-Split; Test type: Other; p < 0.005, t-test, 2 sided — Chicago BPS Total Score -- 1 was lower than 3,4,5; 2 was lower than 5. Modified Chicago BPS Total Score -- 1 were lower than 5. Chicago BPS Fluid Score -- 1 was dryer than 3,4,5; 2 was dryer than 3,4,5; 3 was wetter than 4,5

2. Secondary Outcome: Boston Bowel Preparation Scale
Description: The quality of the colon preparation as graded using Boston Bowel Preparation total scores is range from 0 (very poor) to 9 (outstanding).
Time Frame: At completion of colonoscopy - day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MiraLAX 306 g (Day-Prior) | MiraLAX 357 g (Day-Prior) | MiraLAX 306 g (Split-Dose) | MoviPrep (Split-Dose) | SUPREP (Split-Dose)
Number analyzed (Participants) | 200 | 200 | 200 | 200 | 200
units on a scale | 8.39 (1.36) | 8.57 (1.16) | 8.66 (1.16) | 8.80 (1.04) | 8.80 (0.77)
Statistical Analysis 1: Comparison: MiraLAX 306 g (Day-Prior) vs MiraLAX 357 g (Day-Prior) vs MiraLAX 306 g (Split-Dose) vs MoviPrep (Split-Dose) vs SUPREP (Split-Dose); All 5 arms were compared pair-wise. 1=G+PEG-306 2=G+PEG-357 3=G+PEG-Split 4=PEG+Asc-Split 5=SS-Split; Test type: Other; p < 0.001, t-test, 2 sided — 1 was lower than 4,5

3. Secondary Outcome: Adequate/Inadequate Scale
Description: The cleanliness of the colon as rated by the gastroenterologist using an adequate/inadequate scale where an adequate preparation is defined as being able to see at least 95% of the mucosa of the colon after washing and suctioning; otherwise, the preparation is rated as inadequate.
Time Frame: At completion of colonoscopy - day 1
Measure: Count of Participants; unit: Participants
Arm/Group | MiraLAX 306 g (Day-Prior) | MiraLAX 357 g (Day-Prior) | MiraLAX 306 g (Split-Dose) | MoviPrep (Split-Dose) | SUPREP (Split-Dose)
Number analyzed (Participants) | 200 | 200 | 200 | 200 | 200
Participants
  Adequate | 195 | 196 | 198 | 197 | 197
  Inadequate | 5 | 4 | 2 | 3 | 3
Statistical Analysis 1: Comparison: MiraLAX 306 g (Day-Prior) vs MiraLAX 357 g (Day-Prior) vs MiraLAX 306 g (Split-Dose) vs MoviPrep (Split-Dose) vs SUPREP (Split-Dose); All 5 arms were compared pair-wise; Test type: Other; p > 0.005, Chi-squared

ADVERSE EVENTS:
Arm/Group | MiraLAX 306 g (Day-Prior) | MiraLAX 357 g (Day-Prior) | MiraLAX 306 g (Split-Dose) | MoviPrep (Split-Dose) | SUPREP (Split-Dose)
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200 | 0/200 | 0/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200 | 0/200 | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 119/200 | 122/200 | 126/200 | 110/200 | 111/200
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MiraLAX 306 g (Day-Prior) (N=200) | MiraLAX 357 g (Day-Prior) (N=200) | MiraLAX 306 g (Split-Dose) (N=200) | MoviPrep (Split-Dose) (N=200) | SUPREP (Split-Dose) (N=200)
Nausea (Gastrointestinal disorders) | 65 | 80 | 66 | 65 | 70
Vomiting (Gastrointestinal disorders) | 18 | 23 | 12 | 8 | 13
Abdominal Cramps/Pain (Gastrointestinal disorders) | 66 | 70 | 68 | 75 | 78
Bloating (Gastrointestinal disorders) | 119 | 122 | 126 | 110 | 111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes